CLINICAL TRIAL: NCT00000847
Title: A Phase I Safety and Immunogenicity Trial of Live Recombinant Canarypox ALVAC-HIV (vCP205) and HIV-1 SF-2 rgp120 in HIV-1 Uninfected Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: AVEG 022A; 10573 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; HIV Envelope Protein gp120; AIDS Vaccines; HIV Seronegativity; Avipoxvirus; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: ALVAC-HIV MN120TMG (vCP205)
Biological: ALVAC-RG Rabies Glycoprotein (vCP65)
Biological: rgp120/HIV-1 SF-2

SUMMARY:
To evaluate the safety and immunogenicity of high-titered ALVAC-HIV MN120TMG (vCP205) given sequentially or simultaneously with rgp120/HIV-1SF2 in MF59 adjuvant emulsion in HIV-negative volunteers.

ALVAC-HIV vCP205 is a second-generation candidate vaccine that can be used to induce a humoral and cellular response against several antigens. vCP205 expresses proteins from two strains of HIV (MN and LAI). rgp120/HIV-1SF2 expresses proteins from a different strain of HIV. This study will help to show how the immune system responds to proteins from more than one strain of virus.

DETAILED DESCRIPTION:
ALVAC-HIV vCP205 is a second-generation candidate vaccine that can be used to induce a humoral and cellular response against several antigens. vCP205 expresses proteins from two strains of HIV (MN and LAI). rgp120/HIV-1SF2 expresses proteins from a different strain of HIV. This study will help to show how the immune system responds to proteins from more than one strain of virus.

Six groups of 25 volunteers each are randomized to receive simultaneous or sequential doses of ALVAC-HIV vCP205 and SF2 rgp120 or control vaccines (ALVAC-RG rabies glycoprotein vCP65 or BIOCINE Placebo Vaccine 2). In each group, 21 volunteers receive vaccine and 4 receive control vaccines. Volunteers are stratified by lower or higher risk sexual behavior. Immunizations are given to three groups at months 0, 1, 3, 6, 9, and 12, and to the other three groups at months 0, 1, 6, 9, and 12. Volunteers are followed for 24 months.

ELIGIBILITY:
Inclusion Criteria

Volunteers must have:

* Normal history and physical exam.
* Negative ELISA and Western blot for HIV.
* CD4 count >= 400 cells/mm3.
* Normal urine dipstick with esterase and nitrite.

NOTE:

* No more than 10 percent of volunteers in each stratum may be over age 50.

Risk Behavior:

Allowed for volunteers stratified to the higher risk stratum:

High risk behavior for HIV infection, such as

* injection drug use within the past 12 months.
* higher or intermediate risk sexual behavior.

Exclusion Criteria

Co-existing Condition:

Subjects with the following symptoms or conditions are excluded:

* Positive hepatitis B surface antigen.
* Medical or psychiatric condition (such as recent suicidal ideation or present psychosis) that precludes compliance.
* Occupational responsibilities that preclude compliance.
* Active syphilis. NOTE: Subjects with serology documented to be a false positive or due to a remote (> 6 months) treated infection are eligible.
* Active tuberculosis. NOTE: Subjects with a positive PPD and a normal chest x-ray showing no evidence of TB and not requiring isoniazid therapy are eligible.
* Allergy to egg products or neomycin.
* Occupational exposure to birds.

Subjects with the following prior conditions are excluded:

* History of immunodeficiency, chronic illness, autoimmune disease, or use of immunosuppressive medications.
* History of anaphylaxis or other serious adverse reactions to vaccines.
* Prior immunization against rabies.
* History of serious allergic reaction to any substance, requiring hospitalization or emergent medical care (e.g., Stevens-Johnson syndrome, bronchospasm, or hypotension).
* Prior psychiatric condition (such as history of suicide attempts or past psychosis) that precludes compliance.
* History of cancer unless there has been surgical excision that is considered to have achieved cure.

Prior Medication:

Excluded:

* Live attenuated vaccines within 60 days prior to study entry. NOTE: Medically indicated killed or subunit vaccines (e.g., influenza, pneumococcal) do not exclude if administered at least 2 weeks from HIV immunizations.
* Experimental agents within 30 days prior to study entry.
* Prior HIV vaccines.
* Prior rabies immunization.

Prior Treatment:

Excluded:

* Blood products or immunoglobulin within the past 6 months.

For volunteers stratified to the lower risk stratum:

High risk behavior for HIV infection, such as

* injection drug use within the past 12 months.
* higher or intermediate risk sexual behavior.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150
Dates: Study Completion 1999-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey L, Study Chair
Locations (6):
- United States (6):
  - UAB AVEG, Birmingham, Alabama
  - JHU AVEG, Baltimore, Maryland
  - St. Louis Univ. School of Medicine AVEG, St Louis, Missouri
  - Univ. of Rochester AVEG, Rochester, New York
  - Vanderbilt Univ. Hosp. AVEG, Nashville, Tennessee
  - UW - Seattle AVEG, Seattle, Washington

REFERENCES:
- [Background] Corey L, Weinhold K, Montefiori D, McElrath J, Excler JL, Duliege AM, Stablein D. Combination candidate HIV vaccines using a canarypox vector (vCP205) followed by boosting with gp120(SF-2). Conf Retroviruses Opportunistic Infect. 1997 Jan 22-26;4th:209 (abstract no LB18)
- [Background] Evans T, Corey L, Clements-Mann ML, Weinhold K, Belshe RB, Excler JL, Duliege AM. CD8+ CTL induced in AIDS vaccine evaluation group phase I trials using canarypox vectors (ALVAC) encoding multiple HIV gene products (vCP125, vCP205, vCP300) given with or without subunit boost. Int Conf AIDS. 1998;12:277 (abstract no 495/21192)
- [Background] Corey L, Weinhold K, Montefiori D, Stablein D. CTL and neutralizing antibody responses with a combination HIV-1 vaccine regimen. Int Conf AIDS. 1998;12:636 (abstract no 33221)
- [Background] Kaslow RA, Rivers C, Goepfert P, Tang J, El Habib R, Weinhold K, Mulligan MJ. Association of HLA class I alleles with cytotoxic T-lymphocyte (CTL) responses to gag and env in recipients of ALVAC-HIV canarypox vaccines. 7th Conference on Retroviruses and Opportunistic Infections. 2000 Jan 30-Feb 2 [Poster 818]
- [Background] AIDS Vaccine Evaluation Group 022 Protocol Team. Cellular and humoral immune responses to a canarypox vaccine containing human immunodeficiency virus type 1 Env, Gag, and Pro in combination with rgp120. J Infect Dis. 2001 Feb 15;183(4):563-70. doi: 10.1086/318523. Epub 2001 Jan 18. PMID 11170981
- [Background] Gupta K, Hudgens M, Corey L, McElrath MJ, Weinhold K, Montefiori DC, Gorse GJ, Frey SE, Keefer MC, Evans TG, Dolin R, Schwartz DH, Harro C, Graham B, Spearman PW, Mulligan M, Goepfert P; AIDS Vaccine Evaluation Group. Safety and immunogenicity of a high-titered canarypox vaccine in combination with rgp120 in a diverse population of HIV-1-uninfected adults: AIDS Vaccine Evaluation Group Protocol 022A. J Acquir Immune Defic Syndr. 2002 Mar 1;29(3):254-61. doi: 10.1097/00126334-200203010-00005. PMID 11873074
- [Background] Bender TJ, Tang J, Rivers C, Mulligan MJ, Kaslow RA. Grouping by HLA class I supertype does not enhance HLA associations with CTL responses to ALVAC-HIV canarypox vaccine components. 8th Conf Retro and Opportun Infect. 2001 Feb 4-8 (abstract no 193)